CLINICAL TRIAL: NCT04669964
Title: Evaluating the Efficacy of a Standardized Hydration Protocol After Ileostomy Creation
Brief Title: Evaluating Ileostomy Hydration Protocol
Status: Withdrawn | Type: Observational
Why Stopped: Change in routine care was not implemented at organization
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-73
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Ileostomy - Stoma; Ileostomy; Complications; Dehydration
Keywords: ileostomy; dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High-Risk For Dehydration: Patients with an Ileostomy output of >1L at discharge.
  Interventions: Procedure: Intravenous Hydration

INTERVENTIONS:
Procedure: Intravenous Hydration — Patients will receive daily intravenous hydration of normal saline based on their ileostomy output.

SUMMARY:
This is a prospective observational study on patients who undergo an ileostomy creation after implementing a hydration algorithm as routine care at Robert Packer Hospital. The Department of Surgery will be implementing a protocol to prevent dehydration for patients with high output ileostomies. Patients with high output ileostomies are at an increased risk for readmission for dehydration. By reviewing the data after applying this standardized hydration protocol, we can assess its efficacy on readmission rates and comorbidities stemming from dehydration.

DETAILED DESCRIPTION:
As of January 1, 2021, Robert Packer Hospital will implement a standardized hydration protocol for patients at high risk for readmission due to dehydration.

All postoperative ileostomy patients will be provided the following instructions at the bedside to ensure complete comprehension:

1. Stoma maintenance education
2. Hydration recommendations
3. Intake and Output Worksheet education and trial

The colorectal surgeons standardized the postoperative medical management of ileostomy output.

Before discharge, the healthcare providers will complete a "Discharge Assessment Checklist".

On the day of discharge, patients will be categorized by the "Discharge Algorithm for Patients with Ileostomies." The algorithm will assign patients by their ileostomy output and determine their next management steps.

After discharge, all patients will record their fluid input and output using the "Daily Measurement of Intake/Output Worksheet" which will be used to monitor hydration over time. Patients who are high risk will receive outpatient intravenous hydration therapy. At each intravenous therapy appointment, the health care provider will review the Outpatient Intravenous Hydration Algorithm to determine the volume of fluid to distribute or if re-evaluation is necessary.

Data Collection After starting the standardized hydration protocol, researchers will prospectively collect data from monthly reports of patients who received an ileostomy creation.

Researchers will not mask the patients, care providers, investigators, and outcomes assessors.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age will be eligible for this study.
* Patients who received emergent or elective end or loop ileostomy during the index admission will be eligible for this study.

Exclusion criteria:

- Patients who have not received an ileostomy creation at Robert Packer Hospital will be ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over the age of 18 years of age who received an emergent or elective end or loop ileostomy at Robert Packer Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Readmission with 30 days | 30 days after discharge for ileostomy creation
  Unplanned hospital readmission within 30 days of ileostomy creation. Researchers will determine unplanned hospital readmissions through monthly generated patient reports and validated by chart review.

SECONDARY OUTCOMES:
Readmission | 60 and 90 days after discharge for ileostomy creation
  Unplanned hospital readmission within 60 and 90 days of surgery. Researchers will determine unplanned hospital readmissions through monthly generated patient reports and validated by chart review.
Emergency Department Visits | 30, 60, and 90 days after discharge for ileostomy creation
  Emergency department visits within 30, 60, and 90 days of surgery. Researchers will determine emergency department visits through monthly generated patient reports and validated by chart review.
Dehydration Events | 30, 60, and 90 days after discharge for ileostomy creation
  The number of clinically significant dehydration events within 30, 60, and 90 days of surgery. Researchers will determine the number of clinically significant dehydration events through monthly generated patient reports and validated by chart review.
Reoperation | 30, 60, and 90 days after discharge for ileostomy creation
  The incidence of reoperation within 30, 60, and 90 days of surgery. Researchers will determine the incidence of reoperation through monthly generated patient reports and validated by chart review.
Mortality | 30, 60, and 90 days after discharge for ileostomy creation
  Mortality rates within 30, 60, and 90 days of surgery. Researchers will determine mortality through monthly generated patient reports and validated by chart review

CONTACTS AND LOCATIONS:
Overall Officials: Burt Cagir M FACS, Principal Investigator — Robert Packer Hospital
Locations (1):
- Guthrie Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Murken DR, Bleier JIS. Ostomy-Related Complications. Clin Colon Rectal Surg. 2019 May;32(3):176-182. doi: 10.1055/s-0038-1676995. Epub 2019 Apr 2. PMID 31061647
- [Background] Vergara-Fernandez O, Trejo-Avila M, Santes O, Solorzano-Vicuna D, Salgado-Nesme N. Predictors of dehydration and acute renal failure in patients with diverting loop ileostomy creation after colorectal surgery. World J Clin Cases. 2019 Jul 26;7(14):1805-1813. doi: 10.12998/wjcc.v7.i14.1805. PMID 31417926
- [Background] Ahmad SJ, Khan A, Madhotra R, K Exadaktylos A, Milioto ME, Macfaul G, Rostami K. Semi-elemental diet is effective in managing high output ileostomy; a case report. Gastroenterol Hepatol Bed Bench. 2019 Spring;12(2):169-173. PMID 31191843
- [Background] Al-Mazrou AM, Suradkar K, Mauro CM, Kiran RP. Characterization of Readmission by Day of Rehospitalization After Colorectal Surgery. Dis Colon Rectum. 2017 Feb;60(2):202-212. doi: 10.1097/DCR.0000000000000734. PMID 28059917
- [Background] Abdalla S, Scarpinata R. Early and Late Closure of Loop Ileostomies: A Retrospective Comparative Outcomes Analysis. Ostomy Wound Manage. 2018 Dec;64(12):30-35. PMID 30516478
- [Background] van Loon YT, Poylin VY, Nagle D, Zimmerman DDE. Effectiveness of the Ileostomy Pathway in Reducing Readmissions for Dehydration: Does It Stand the Test of Time? Dis Colon Rectum. 2020 Aug;63(8):1151-1155. doi: 10.1097/DCR.0000000000001627. PMID 32692076
- [Background] Nagle D, Pare T, Keenan E, Marcet K, Tizio S, Poylin V. Ileostomy pathway virtually eliminates readmissions for dehydration in new ostomates. Dis Colon Rectum. 2012 Dec;55(12):1266-72. doi: 10.1097/DCR.0b013e31827080c1. PMID 23135585
- [Background] Grass F, Lovely JK, Crippa J, Hubner M, Mathis KL, Larson DW. Potential Association Between Perioperative Fluid Management and Occurrence of Postoperative Ileus. Dis Colon Rectum. 2020 Jan;63(1):68-74. doi: 10.1097/DCR.0000000000001522. PMID 31633601
- [Background] Kristensen K, Qvist N. The Acute Effect of Loperamide on Ileostomy Output: A Randomized, Double-Blinded, Placebo-Controlled, Crossover Study. Basic Clin Pharmacol Toxicol. 2017 Dec;121(6):493-498. doi: 10.1111/bcpt.12830. Epub 2017 Jul 10. PMID 28627732
- [Background] Parli SE, Pfeifer C, Oyler DR, Magnuson B, Procter LD. Redefining "bowel regimen": Pharmacologic strategies and nutritional considerations in the management of small bowel fistulas. Am J Surg. 2018 Aug;216(2):351-358. doi: 10.1016/j.amjsurg.2018.01.040. Epub 2018 Feb 12. PMID 29448989
- [Background] Bleier JI, Hedrick T. Metabolic support of the enterocutaneous fistula patient. Clin Colon Rectal Surg. 2010 Sep;23(3):142-8. doi: 10.1055/s-0030-1262981. PMID 21886463
- See also: Study from the Agency for Healthcare Research and Quality estimated that the mean cost per readmission for ileostomy procedures is $15,434 — https://hcup-us.ahrq.gov/reports/statbriefs/sb153.jsp